CLINICAL TRIAL: NCT00261222
Title: Efficacy of Amodiaquine in the Treatment of Uncomplicated Falciparum Malaria in Young Children of Burkina Faso
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFB544-A8-AQ2005
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2006-10

CONDITIONS: Malaria
Keywords: Amodiaquine; Efficacy; Malaria; Burkina Faso
MeSH Terms: conditions — Malaria | interventions — Amodiaquine

INTERVENTIONS:
Drug: Amodiaquine

SUMMARY:
Design: Single-centre

Indication: Malaria caused by Plasmodium falciparum Objectives: To determine and compare the efficacy of AQ treatment in young children with uncomplicated falciparum malaria in the rural and the urban study area of the Centre de Recherche en Santé de Nouna (CRSN).

Population: Children aged 6-59 months with uncomplicated falciparum malaria (axillary temperature ≥ 37.5°C + ≥ 2.000 P. falciparum asexual parasites per µl blood) from the health centre situated in the villages of Bagala, Bourasso and Kemena and from Nouna town hospital outpatient department.

Sample size: N=120

Treatment: All children will receive a total dose of 25 mg/kg oral AQ over a period of three days (first and second day: 10mg/kg, third day: 5mg/kg).

Statistical procedures: The primary analysis parameter is the proportion of clinical failures on day 14. Secondary parameters are the rate of clinical failures on day 28 (with and without PCR correction), the rate of early clinical failures, the rate of late parasitological failures (day 14 and day 28), and the rate of adverse events. Data will be analysed in the overall group of study children and for rural (n=50) and urban (n=50) study children separately.

Study duration and dates: The study will be implemented in September-December 2005.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-59 months
* Uncomplicated falciparum malaria (axillary temperature ≥ 37.5°C and ≥ 2.000 P. falciparum asexual parasites per µl blood)
* Written informed consent given by the parents/caretakers

Exclusion Criteria:

* Complicated or severe malaria (repeated vomiting, seizures or other neurological impairment, haemoglobin < 7 g/dl or haematocrit < 21%)
* Any apparent significant disease (e. g. pneumonia, meningitis, hepatitis, severe diarrhoea, measles, severe malnutrition)
* Malaria treatment with western drugs and/or antibiotics with anti malarial potency during last 7 days except chloroquine.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 2005-09; Study Completion 2005-11

PRIMARY OUTCOMES:
Total clinical failure rate on day 14.
Clinical failure rate on day 14 in rural study area.
Clinical failure rate on day 14 in urban study area.

SECONDARY OUTCOMES:
Total clinical failure rate on day 28.
Clinical failure rate on day 28 in rural study area.
Clinical failure rate on day 28 in urban study area.
Total early clinical failure rate.
Early clinical failure rate in rural study area.
Early clinical failure rate in urban study area.
Total late parasitological failure rate on day 14 and 28.
Late parasitological failure rate on day 14 and 28 in rural study area.
Late parasitological failure rate on day 14 and 28 in urban study area.
Incidence of observed and self-reported adverse events over the 28 days observation period
Monitoring of concomitant drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Germain Mandi, MD, Principal Investigator — Centre de Recherche en Santé de Nouna; Olaf Mueller, MD, PhD, Study Director — University of Heidelberg, Germany, Institute of Tropical Medecine and Public Health
Locations (1):
- Centre de Recherche en Santé de Nouna (CRSN), Nouna, Burkina Faso